CLINICAL TRIAL: NCT03606018
Title: A Randomized Duble Blinded Two-way Crossover Single-dose Pharmacokinetics and Pharmacodynamics Study of Insulin Lispro Mix 25 (LLC "GEROPHARM", Russia) Versus Humalog® Mix 25 (Eli Lilly) in Healthy Subjects Using the Euglycemic Clamp Technique
Brief Title: A Study to Compare Pharmacokinetics and Pharmacodynamics of Insulin Lispro Mix 25 to Humalog® Mix 25 in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LISPRO-25-CL
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Clamp Study
Keywords: Pharmacokinetics; Pharmacodynamics; Insulin Lispro

STUDY DESIGN:
Intervention Model Description: two-way crossover
Who Masked: Outcomes Assessor
Masking Description: This study was blinded for Sponsor, investigators and analytical laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Lispro Mix 25 (Experimental): Single subcutaneous administration of Insulin Lispro Mix 25 in dose 0.4 IU / kg
  Interventions: Drug: Insulin Lispro Mix 25
- Humalog® Mix 25 (Active Comparator): Single subcutaneous administration of Humalog® Mix 25 in dose 0.4 IU / kg
  Interventions: Drug: Humalog® Mix 25

INTERVENTIONS:
Drug: Insulin Lispro Mix 25 — insulin lispro biphasic in doses 0.4 ME/kg
  Other Names: insulin lispro biphasic
  Arms: Insulin Lispro Mix 25
Drug: Humalog® Mix 25 — insulin lispro biphasic in doses 0.4 ME/kg
  Other Names: insulin lispro biphasic
  Arms: Humalog® Mix 25

SUMMARY:
Pharmacokinetics and pharmacodynamics study Study of 2 formulation of insulin lispro mix 25 (Insulin Lispro Mix 25 GEROPHARM vers. Humalog® Mix 25 Eli Lilly)

DETAILED DESCRIPTION:
A randomized duble blinded two-way crossover single-dose pharmacokinetics and pharmacodynamics study of Insulin Lispro Mix 25 (LLC "GEROPHARM", Russia) versus Humalog® Mix 25 (Eli Lilly) in normal healthy subjects using the euglycemic clamp technique

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Caucasian males having a confirmed healthy diagnosis as per data of standard clinical, laboratory, and instrumental examination methods.
3. Age of 18-50 (both incl.).
4. Body mass index equal to 18.5-27.0 kg/m2.
5. Volunteers' consent to all restrictions imposed during the study, including adequate methods of contraception.

Exclusion Criteria:

1. Acute inflammatory diseases within 3 weeks before the screening period
2. Episodes of hypoglycemia in the anamnesis, or the presence in the family history of cases of a verified diagnosis of diabetes mellitus in the immediate family
3. Fasting plasma glucose> 6.1 mmol / L
4. HbA1C> 6%
5. Oral glucose tolerance test - blood glucose level ≥ 7.8 mmol / l (2 hours after loading with glucose)
6. Deep vein thrombosis of lower extremities in a history of life or in a family history.
7. Nicotine dependence (use of tobacco less than 6 months before the start of screening)
8. Taking medications, phytopreparations, biologically active supplements less than 14 days before screening
9. Receiving more than 10 units. alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of wine or 50 ml of strong alcohol) or anamnestic information about alcoholism.
10. Donor blood donation in excess of 450 ml, less than 2 months before the study.
11. Participation in a clinical trial of any medications less than 3 months before the start of screening
12. Positive test results for hepatitis C or hepatitis B, HIV, syphilis.
13. Anamnesis information about drug and / or drug dependence and / or substance abuse.
14. Positive test for alcohol content in the exhaled air.
15. A positive test for the content of drugs in the urine.
16. Presence of suspicions of an inflammatory disease of the urinary system as a result of urinalysis.
17. Presence of mental illnesses in the anamnesis.
18. Mental, physical and other reasons that do not allow to adequately assess their behavior and properly fulfill the conditions of the research protocol.
19. Any other conditions that make it difficult, according to the informed opinion of the investigating physician, that volunteer participation in studies
20. Increased sensitivity in the history of heparin, insulin or any of the excipients of the study drugs
21. Weighed allergic anamnesis
22. Abnormalities of the ECG and laboratory parameters from the norms
23. Deviations in basic vital signs: systolic blood pressure is below 100 mm Hg. or above 130 mm Hg, the diastolic blood pressure is below 70 mm Hg. or above 90 mm Hg; heart rate less than 60 or greater than 80
24. Deviations in basic vital signs: systolic blood pressure <100 mmHg. or> 130 mm Hg, diastolic blood pressure <70 mm Hg. Art. or> 90 mm Hg. Art. heart rate <60 or> 80 per minute.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In women of childbearing age, the cyclicity of the hormonal status may affect insulin sensitivity at different stages of the study. Therefore, to exclude the influence of the cyclicity factor of the menstrual period on insulin sensitivity in women, only males have been included in the this study
Enrollment: 48 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Cmax | -0.5, 0 hour (pre-dose) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5, 14 hour post-dose
  Pharmacokinetics of insulin lispro by Assessment of Observed Maximum Plasma Concentration (Cmax)
AUC(0-t) | -0.5, 0 hour (pre-dose) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 5.75, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5, 14 hour post-dose
  Pharmacokinetics of insulin Lispro by Assessment of Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t))

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - FSBI"ENDOCRINOLOGY NMRC" Ministry of Health of the Russian Federation, Moscow
  - LLL "BioEq", Saint Petersburg